CLINICAL TRIAL: NCT01492114
Title: Double-blind Cross-over Randomised Controlled Trial on the Anti-inflammatory and Antioxidant Effects of Resveratrol on Healthy Adults.
Brief Title: Anti-inflammatory and Antioxidant Effects of Resveratrol on Healthy Adults.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Simona Bo, MD, Department of Internal Medicine, University of Turin, Italy
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: sbo2011
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Subclinic Inflammation; Redox Status
Keywords: C-reactive protein; Resveratrol; Redox index
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resveratrol first (Experimental): Subjects in the group "resveratrol first" will be submitted to: 30 days of treatment with Transmax (resveratrol, 500 mg, Biotivia Bioceuticals LLC), one tablet/day in the morning at fasting; then to 30 days of wash-out (no supplementation), and then to 30 days of treatment with placebo (one tablet/day in the morning at fasting).
  Interventions: Dietary Supplement: Resveratrol
- Placebo first (Active Comparator): Subjects in the group "Placebo first" will be submitted to: 30 days of treatment with placebo, one tablet/day in the morning at fasting; than to 30 days of wash-out (no supplementation), and then to 30 days of treatment with Transmax (resveratrol, 500 mg) (one tablet/day in the morning at fasting).
  Interventions: Dietary Supplement: resveratrol

INTERVENTIONS:
Dietary Supplement: Resveratrol — Subjects in the group "resvetarol first" will be submitted to: 30 days of treatment with Transmax (resveratrol, 500 mg, Biotivia Bioceuticals LLC), one tablet/day in the morning at fasting; then to 30 days of wash-out (no supplementation), and then to 30 days of treatment with placebo (one tablet/day in the morning at fasting).
  Arms: Resveratrol first
Dietary Supplement: resveratrol — Subjects in the group "Placebo first" will be submitted to: 30 days of treatment with placebo, one tablet/day in the morning at fasting; than to 30 days of wash-out (no supplementation), and then to 30 days of treatment with Transmax (resveratrol, 500 mg) (one tablet/day in the morning at fasting).
  Arms: Placebo first

SUMMARY:
This research will investigate the hypothesis that resveratrol when given orally to healthy adult smokers induces a decrease in the inflammatory and oxidative mediators which characterize the low-grade systemic inflammatory state and the oxidants-antioxidants imbalance of tobacco users.

DETAILED DESCRIPTION:
The effect of resveratrol in humans is still not well defined. The number of studies on resveratrol has increased extraordinarily since 1997, when its anticancer effect has been reported. However, most of these studies are in-vitro or animal studies. Preclinical observations in humans suggest that resveratrol is safe and has potential in the treatment of obesity and insulin resistance in humans.

In particular, it improves insulin sensitivity, which might be due to a resveratrol-induced decrease in oxidative stress that leads to a more efficient insulin signalling via the Akt pathway. Studies on toxicity of resveratrol in humans demonstrated that this compound is well tolerated and no adverse effect has been found with higher dosage (5g/day). Resveratrol is available to people over-the-counter in health food stores and the internet as a dietary supplement. In humans, resveratrol is efficiently absorbed after oral administration; however, rapid phase II metabolism drastically limits its plasma bio-availability. The high concentrations of resveratrol in colorectal tissues, in excess of that required for activity in vitro, supports the colon as a target organ. The efficacy of resveratrol in other tissues may be largely dependent on whether its metabolites have significant activity or are able to regenerate resveratrol either locally or systemically (e.g. some metabolites, mainly sulfate-conjugated resveratrol, show biological effects in cellular models).

There are only a few studies evaluating the anti-inflammatory properties of resveratrol in humans. An extract of Polygonum Cuspidatum containing resveratrol given for 6-weeks to 10 healthy subjects was able to significantly suppress plasma concentrations of inflammatory cytokines (C-reactive protein, interleukin-6, tumor necrosis factor-α). Similarly, a nutritional supplement containing resveratrol plays an acute antioxidant and antiinflammatory effects in the postprandial state after a high-fat, high-carbohydrate meal in 10 healthy females.

The anti-inflammatory and antioxidant effects of resveratrol may be particularly interesting for smokers. Resveratrol increases the NO bioavailability and the inhibition of cyclooxygenase and 5-lipoxygenase activity of Cox-1 and it prevents the vascular leucocyte migration into damaged organs by decreasing the expression of endothelial vascular adhesion molecules and of pro-inflammatory genes. The inflammatory responses induced by oxidized LDL (low-density lipoproteins) are partially avoided by the addition of reveratrol and the authors concluded that it could affect vascular inflammation or/and injury not only as antioxidant, but also as modulator of inflammatory redox signalling pathways.

However, there are currently no published demonstrations of therapeutic or protective effects of resveratrol in appropriately designed clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* age 20-50 years
* actual smoking (≥5 cigarettes/die)
* mean alcohol consumption <30g/day
* absence of known hyperglycaemia, hypertension, cardiovascular disease, impaired renal function, liver disease, or any other systemic conditions -no use of any drug -oestrogen excluded-
* not being on a particular diet and/or vitamin or other nutrient or integrator supplementation during the least 6-months

Exclusion Criteria:

* actual pregnancy -known hyperglycaemia, hypertension, cardiovascular disease, impaired renal function, liver disease, or any other systemic chronic or acute conditions, use of any drug -oestrogen excluded-
* being on a particular diet and/or vitamin or other nutrient or integrator supplementation during the last six months
* mean alcohol consumption ≥30g/day
* body mass index (BMI)>30 kg/m2
* subject unable to give his/her informed consent.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
C-reactive protein | At baseline and every 30 days for three months
  To evaluate before-after changes in circulating concentrations of C-reactive protein (CRP), an inflammation marker, in smokers submitted to resveratrol supplementation when compared to smokers treated with placebo

SECONDARY OUTCOMES:
TAS (total antioxidant status) | At baseline and every 30-days for three months
  To evaluate before-after changes in circulating fasting concentrations of the following parameters:
  -markers of oxidative stress: TAS (total antioxidant status.
4-hydroxynonenal | At baseline and after 30-days for three months
  To evaluate before-after changes in circulating fasting concentrations of the following parameters:
  -markers of oxidative stress: 4-hydroxynonenal
nitrotyrosine | At baseline and every 30-days for three months
  To evaluate before-after changes in circulating fasting concentrations of the following parameters:
  -markers of oxidative stress: nitrotyrosine.
endothelial nitric oxide synthase (eNOS)-polymorphism | At baseline and every 30-days for three months
  To evaluate before-after changes in circulating fasting concentrations of the following parameters:
  -markers of oxidative stress: endothelial nitric oxide synthase (eNOS)-polymorphism
superoxide dismutase (SOD2)-polymorphism | At baseline and every 30-days for three months
  To evaluate before-after changes in circulating fasting concentrations of the following parameters:
  -markers of oxidative stress: superoxide dismutase (SOD2)-polymorphism.
catalase-polymorphism | At baseline and every 30-days for three months
  To evaluate before-after changes in circulating fasting concentrations of the following parameters:
  -markers of oxidative stress: catalase-polymorphism
interleukin-6 | At baseline and every 30-days for three months
  To evaluate before-after changes in circulating fasting concentrations of the following parameters:
  -other markers of inflammation: interleukin-6.
pentraxin 3 | At baseline and every 30-days for three months
  To evaluate before-after changes in circulating fasting concentrations of the following parameters:
  -other markers of inflammation: pentraxin 3.
tumor necrosis factor-α | At baseline and every 30-days for three months
  To evaluate before-after changes in circulating fasting concentrations of the following parameters:
  -other markers of inflammation: tumor necrosis factor-α.

CONTACTS AND LOCATIONS:
Overall Officials: Simona Bo, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- Simona Bo, Turin, Turin, Italy